CLINICAL TRIAL: NCT02101697
Title: Reducing AIDS Stigma Among Health Professionals in India
Acronym: DRISTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R01MH093257 (NIH); R01MH093257 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-02 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Stigmatization
Keywords: reduce; Indian health providers
MeSH Terms: conditions — Stereotyping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV Stigma Reduction Intervention (Experimental): The HIV stigma reduction arm group will participate in a promising intervention designed to reduce HIV stigma among health professionals. The intervention builds on results of our previous research, identifying prevalence and drivers of stigma and discrimination in Indian healthcare settings among PLHIV, health care providers, and uninfected patients.The HIV stigma reduction intervention consists of two computer-administered sessions and one group session.
  Interventions: Behavioral: HIV Stigma Reduction Intervention
- Time Matched Control Group (Placebo Comparator): The time-matched control group will also receive three sessions; two administered by computers and one in small group format to control for attention effects. However, rather than AIDS stigma, the content will be focused on diabetes management (a disease not considered to be stigmatized).
  Interventions: Behavioral: HIV Stigma Reduction Intervention

INTERVENTIONS:
Behavioral: HIV Stigma Reduction Intervention — The HIV stigma reduction intervention consists of two computer-administered sessions and one group session.
  Session 1. (approx. 60 min). Introduction of the concepts of stigma and discrimination, vulnerable populations and symbolic stigma delivered in an interactive tablet format, using games and videos.
  Session 2. (approx. 60 min). Interactive activities to address HIV transmission myths and misconceptions and the importance of universal precautions.
  Session 3. (approx 90 min). Patient interaction skills. In person interactive group session co-facilitated by PLHIV and staff focusing on skills building through role-plays and feedback.
  Our previous research has found that these modules address factors identified as contributing to health professionals' stigma.

SUMMARY:
This Randomized Controlled Trial has been designed to test the efficacy of a behavioral intervention to reduce HIV-related stigma among nursing students and ward attendants in 16 sites in South India and 8 sites in North India.

DETAILED DESCRIPTION:
Across the globe, HIV stigma inflicts hardship and suffering on people with HIV and has been found to reduce the likelihood of seeking HIV counseling and testing and PMTCT. Stigma also deters infected individuals from disclosing their status, seeking timely medical treatment for HIV-related problems, reduces ART adherence, and leads to delays in clinic appointments and prescription refills, which can lead to virologic failure and the development and transmission of drug resistance. Medical professionals unfortunately constitute a significant source of stigma for PLHIV.

This study will evaluate the efficacy of a promising intervention designed to reduce HIV stigma among Indian health professionals. The intervention builds on results of our previous research, identifying prevalence and drivers of stigma and discrimination in Indian healthcare settings among PLHIV, health care providers and uninfected patients.

Specifically, the study will:

1. Adapt our pilot-tested 3-session stigma reduction intervention for partial tablet-based delivery to increase its long-term sustainability in health care settings. The two tablet-administered sessions of the intervention use interactive touch screen methodology and video vignettes tailored to situations likely to be encountered by Indian nurses and ward attendants. The third session focuses on skills-building in a group format and is co-facilitated by a PLHIV.
2. Evaluate the efficacy of the intervention in 24 hospitals in North and South India on:

   1. behavioral manifestations of HIV stigma, including endorsement of coercive policies, behavioral intentions to discriminate, and non/stigmatizing provider-patient interactions.
   2. the factors underlying stigma proposed by our conceptual model and targeted in the intervention modules, including fears and misconceptions regarding casual transmission (instrumental stigma), and negative attitudes toward marginalized, vulnerable groups (symbolic stigma).

ELIGIBILITY:
Inclusion Criteria:

For Nursing Students:

1. being enrolled as a 2nd year nursing student in one of the study colleges,
2. being 18 years or older,
3. being able and willing to participate in the intervention and all assessments.

For ward attendants:

1. having worked as ward attendant at one of the study hospitals for at least a year
2. being 18 years or older,
3. being able and willing to participate in the intervention and all assessments.

Exclusion Criteria:

a) Unwilling or unable to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3733 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
behavioral manifestations of HIV-related stigma | one year
  Evaluate the efficacy of the intervention in a RCT, among nursing students and ward attendants on behavioral manifestations of AIDS stigma including their endorsement of coercive policies, behavioral intentions to discriminate, and non/stigmatizing provider-patient interactions, using face-to-face interviews, computer-based assessments, and ratings by behavioral observers at pre-, 6- and 12 month follow-up.
instrumental and symbolic stigma | one year
  Evaluate the efficacy of the intervention in a RCT, among nursing students and ward attendants on the factors underlying stigma proposed by our conceptual model and targeted in the intervention modules, including fears and misconceptions regarding casual transmission (instrumental stigma), and negative attitudes toward marginalized, vulnerable groups (symbolic stigma), which have consistently been found to drive the behavioral manifestations of AIDS stigma and discrimination.

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Ekstrand, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- St. John's Research Institute/St John's Medical College & Hospital, Bangalore, Karnataka, India

REFERENCES:
- [Background] Shah SM, Heylen E, Srinivasan K, Perumpil S, Ekstrand ML. Reducing HIV stigma among nursing students: a brief intervention. West J Nurs Res. 2014 Nov;36(10):1323-37. doi: 10.1177/0193945914523685. Epub 2014 Feb 25. PMID 24569699
- [Background] Ekstrand ML, Ramakrishna J, Bharat S, Heylen E. Prevalence and drivers of HIV stigma among health providers in urban India: implications for interventions. J Int AIDS Soc. 2013 Nov 13;16(3 Suppl 2):18717. doi: 10.7448/IAS.16.3.18717. PMID 24242265
- [Background] Steward WT, Bharat S, Ramakrishna J, Heylen E, Ekstrand ML. Stigma is associated with delays in seeking care among HIV-infected people in India. J Int Assoc Provid AIDS Care. 2013 Mar-Apr;12(2):103-9. doi: 10.1177/1545109711432315. Epub 2012 Jan 26. PMID 22282878
- [Background] Steward WT, Chandy S, Singh G, Panicker ST, Osmand TA, Heylen E, Ekstrand ML. Depression is not an inevitable outcome of disclosure avoidance: HIV stigma and mental health in a cohort of HIV-infected individuals from Southern India. Psychol Health Med. 2011 Jan;16(1):74-85. doi: 10.1080/13548506.2010.521568. PMID 21218366
- [Background] Nyblade L, Jain A, Benkirane M, Li L, Lohiniva AL, McLean R, Turan JM, Varas-Diaz N, Cintron-Bou F, Guan J, Kwena Z, Thomas W. A brief, standardized tool for measuring HIV-related stigma among health facility staff: results of field testing in China, Dominica, Egypt, Kenya, Puerto Rico and St. Christopher & Nevis. J Int AIDS Soc. 2013 Nov 13;16(3 Suppl 2):18718. doi: 10.7448/IAS.16.3.18718. PMID 24242266
- [Background] Nyblade L, Stangl A, Weiss E, Ashburn K. Combating HIV stigma in health care settings: what works? J Int AIDS Soc. 2009 Aug 6;12:15. doi: 10.1186/1758-2652-12-15. PMID 19660113
- [Background] Varas-Diaz N, Marzan-Rodriguez M. The emotional aspect of AIDS stigma among health professionals in Puerto Rico. AIDS Care. 2007 Nov;19(10):1247-57. doi: 10.1080/09540120701405403. PMID 18071968
- [Background] Varas-Diaz N, Neilands TB. Development and validation of a culturally appropriate HIV/AIDS Stigma Scale for Puerto Rican health professionals in training. AIDS Care. 2009 Oct;21(10):1259-70. doi: 10.1080/09540120902804297. PMID 20024702
- [Background] Ekstrand ML, Bharat S, Ramakrishna J, Heylen E. Blame, symbolic stigma and HIV misconceptions are associated with support for coercive measures in urban India. AIDS Behav. 2012 Apr;16(3):700-10. doi: 10.1007/s10461-011-9888-z. PMID 21290175
- [Background] Li L, Liang LJ, Lin C, Wu Z, Wen Y. Individual attitudes and perceived social norms: Reports on HIV/AIDS-related stigma among service providers in China. Int J Psychol. 2009 Dec;44(6):443-50. doi: 10.1080/00207590802644774. PMID 20090857
- [Background] Li L, Lin C, Wu Z, Wu S, Rotheram-Borus MJ, Detels R, Jia M. Stigmatization and shame: consequences of caring for HIV/AIDS patients in China. AIDS Care. 2007 Feb;19(2):258-63. doi: 10.1080/09540120600828473. PMID 17364408
- [Background] Li L, Wu Z, Wu S, Zhaoc Y, Jia M, Yan Z. HIV-related stigma in health care settings: a survey of service providers in China. AIDS Patient Care STDS. 2007 Oct;21(10):753-62. doi: 10.1089/apc.2006.0219. PMID 17949274
- [Background] Li L, Wu Z, Zhao Y, Lin C, Detels R, Wu S. Using case vignettes to measure HIV-related stigma among health professionals in China. Int J Epidemiol. 2007 Feb;36(1):178-84. doi: 10.1093/ije/dyl256. Epub 2006 Dec 14. PMID 17175545
- [Background] Bharat S. Facing the HIV / AIDS challenge: a study on household and community responses. Health Millions. 1998 Jan-Feb;24(1):15-6, 19. PMID 12348525
- [Background] Mahendra VS, Gilborn L, Bharat S, Mudoi R, Gupta I, George B, Samson L, Daly C, Pulerwitz J. Understanding and measuring AIDS-related stigma in health care settings: a developing country perspective. SAHARA J. 2007 Aug;4(2):616-25. doi: 10.1080/17290376.2007.9724883. PMID 18071613
- [Background] Noar SM, Black HG, Pierce LB. Efficacy of computer technology-based HIV prevention interventions: a meta-analysis. AIDS. 2009 Jan 2;23(1):107-15. doi: 10.1097/QAD.0b013e32831c5500. PMID 19050392
- [Background] Lightfoot M, Rotheram-Borus MJ, Comulada WS, Reddy VS, Duan N. Efficacy of brief interventions in clinical care settings for persons living with HIV. J Acquir Immune Defic Syndr. 2010 Mar;53(3):348-56. doi: 10.1097/QAI.0b013e3181c429b3. PMID 19996978